CLINICAL TRIAL: NCT03365141
Title: Efficacy of Intralesional Triamcinolone Injection in the Treatment of Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Jung Min Bae, Assistant Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VC17MESI0190
Record Dates: First submitted 2017-11-30; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Vitiligo; Treatment; Intralesional Injection; Corticosteroid
Keywords: vitiligo; intralesional injection; corticosteroid; triamcinolone
MeSH Terms: conditions — Vitiligo | interventions — Triamcinolone Acetonide; Phototherapy; Lasers, Excimer; Tacrolimus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): All lesions will treated with NBUVB or excimer laser weekly and application of topical tacrolimus ointment twice daily for a total of 12-week period.
  Intervention: Intralesional injection of triamcinolone acetonide (0.4mg/cc) will be performed weekly.
  Interventions: Drug: Triamcinolone acetonide 0.4mg/cc; Device: Phototherapy (NBUVB or excimer laser); Drug: Topical tacrolimus
- Control group (Active Comparator): All lesions will treated with NBUVB or excimer laser weekly and application of topical tacrolimus ointment twice daily for a total of 12-week period.
  Interventions: Device: Phototherapy (NBUVB or excimer laser); Drug: Topical tacrolimus

INTERVENTIONS:
Drug: Triamcinolone acetonide 0.4mg/cc — * Intralesional injection of dilute triamcinolone acetonide with 2% lidocaine (400mg/20 mL) would be performed to reduce pain when injecting the drug.
  * Once weekly, for a total of 12 weeks
  Arms: Experimental group
Device: Phototherapy (NBUVB or excimer laser) — NBUVB or excimer laser treatment weekly
Drug: Topical tacrolimus — Application of topical tacrolimus ointment twice a day

SUMMARY:
A randomized split-body pilot study was planned to confirm efficacy of intralesiona triamcinolone injection in patients with vitiligo

DETAILED DESCRIPTION:
Intralesional corticosteroid injections have been a long-standing treatment for refractory vitiligo, with some patients showing significant improvement without surgical intervention.

The investigators will perform a randomized split-body pilot trial to test the exact efficacy of intralesional triamcinolone injections. The paired symmetric vitiliginous lesions will be randomized to either control or injection groups. All lesions will be treated with narrowband UV-B phototerapy or excimer laser weekly and twice daily application of topical tacrolimus ointment for a total of 12-week period. Intralesional injections of 0.4mg/cc triamcinolone once a week are given to the experimental group. The degree of repigmentation will be assessed as % from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age : 19 or older
2. A patient who voluntarily agreed to participate in the study by listening to the explanation of the purpose and method of the study
3. A patient who has bilateral two or more vitiligo lesions with similar degree of progression in the face or trunk
4. A patient who has no further response to excimer laser or short wavelength ultraviolet B therapy, which is a conventional treatment for vitiligo

Exclusion Criteria:

1. Patients under the age of 19
2. Patients with enlarged or spreading lesions of vitiligo
3. Patients who do not want to do so or who refuse to write a consent form
4. Patients who are inadequate for triamcinolone acetonide administration (pregnant women, infectious and systemic fungal infections without effective antimicrobial agents, immunosuppression, hypersensitivity reactions to and concomitant use of triamcinolone or its components, spontaneous thrombocytopenia, purpura, herpes simplex, shingles, chicken pox patients)
5. Others those who are deemed unsuitable for the examination at the discretion of the examiner

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-09-15 (Estimated); Study Completion 2018-09-15 (Estimated)

PRIMARY OUTCOMES:
The repigmentation rate (change from baseline) of the vitiliginous patch | Baseline and 12 weeks
  The degree of repigmentation will be assessed as % from baseline by using a computer program.

SECONDARY OUTCOMES:
The adverse effects | every weeks up to 13 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- St. Vincent's Hospital, Suwon, Gyonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No